CLINICAL TRIAL: NCT07197866
Title: An Open-Label Extension, Multi-Centered, Phase 2 Trial to Describe the Safety and Efficacy of TEV-56286 (Emrusolmin) in Participants With Multiple System Atrophy
Brief Title: An Extension Trial to Test if TEV-56286 is Effective in Relieving Multiple System Atrophy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D LLC (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TV56286-NDG-20041; 2025-521642-14-00 (EU CTIS Number)
Record Dates: First submitted 2025-09-26; First posted 2025-09-29 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Multiple System Atrophy
MeSH Terms: conditions — Multiple System Atrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TEV-56286 (Experimental)
  Interventions: Drug: TEV-56286

INTERVENTIONS:
Drug: TEV-56286 — administered orally
  Other Names: Emrusolmin

SUMMARY:
The primary objective of the trial is to describe the long-term safety and tolerability of TEV-56286 administered orally for the treatment of adult participants with Multiple System Atrophy (MSA).

A secondary objective of the trial is to further describe the safety and tolerability of TEV-56286.

The planned total duration of the trial is approximately 100 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Completion of the treatment period and the week 48(V9) visit of the double-blind trial (TV56286-NDG-20039) whilst remaining compliant with trial requirements
* Females of childbearing potential may be included only if they have a negative pregnancy test at the baseline visit
* Females of childbearing potential whose male partners are potentially fertile (ie, no vasectomy) must use highly effective birth control methods for the duration of the trial and for 28 days after the last does of IMP
* Males who are potentially fertile/reproductively competent (not surgically [eg, vasectomy] or congenitally sterile) and their female partners who are of childbearing potential must use, together with their female partners, highly effective birth control methods for the duration of the trial and for 28 days after the last dose of investigational medicinal product

NOTE - Additional criteria apply, please contact the investigator for more information

Exclusion Criteria:

* Is a female participant who is pregnant, plans to become pregnant, or is breastfeeding during the trial
* Is of a vulnerable population (eg, people kept in detention or jail)
* Is using or consuming any prohibited concomitant medications within the specified exclusionary windows of this trial

Note - Additional criteria apply, please contact the investigator for more information

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-09-30 (Actual); Primary Completion 2029-05-03 (Estimated); Study Completion 2029-05-17 (Estimated)

PRIMARY OUTCOMES:
Number of participants experiencing an adverse event | Baseline to Week 100
Number of participants who withdrew from the trial due to an adverse event | Baseline to Week 100

SECONDARY OUTCOMES:
Number of participants with potentially clinically significant vital sign values | Baseline to Week 96
Number of participants with potentially clinically significant laboratory test values (hematology and chemistry) | Baseline to Week 96
Number of participants with potentially clinically significant 12-lead ECG measurements | Baseline to Week 96

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D LLC
Locations (2):
- United States (2):
  - Teva Investigational Site 15544, Boca Raton, Florida
  - Teva Investigational Site 15543, Spokane, Washington

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the study protocol and the statistical analysis plan. Requests will be assessed for scientific merit, product approval status, and conflicts of interest. If the request is approved, patient level data will be de-identified and study documents will be redacted to protect the privacy of trial participants and to protect commercially confidential information. Please email USMedInfo@tevapharm.com to make your request.